CLINICAL TRIAL: NCT01284166
Title: Safety and Efficacy of Triple Combination Therapy With Dorzolamide Hydrochloride / Brimonidine Tartrate / Timolol Ophthalmic Solution in Patients With Glaucoma or Ocular Hypertension
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was never initiated due to company decision. No study subjects were ever enrolled or treated.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dorzo-Brimo-Timo/2010
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — dorzolamide; Brimonidine Tartrate; Timolol; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triple Combination Therapy (Experimental): Triple Combination Therapy with dorzolamide hydrochloride/brimonidine tartrate/timolol ophthalmic solution. One drop of Triple Combination Therapy administered to each eye, twice daily for 12 weeks.
  Interventions: Drug: dorzolamide hydrochloride 2.0%/brimonidine tartrate 0.2%/timolol 0.5% ophthalmic solution

INTERVENTIONS:
Drug: dorzolamide hydrochloride 2.0%/brimonidine tartrate 0.2%/timolol 0.5% ophthalmic solution — 1 drop of Triple Combination Therapy (dorzolamide hydrochloride 2.0%/brimonidine tartrate 0.2%/timolol 0.5% ophthalmic solution) administered to each eye, twice daily for 12 weeks.

SUMMARY:
This study will investigate the safety and efficacy of Triple Combination Therapy with dorzolamide hydrochloride/brimonidine tartrate/timolol ophthalmic solution in patients with glaucoma or ocular hypertension who have elevated IOP on dorzolamide hydrochloride/timolol maleate combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ocular hypertension or glaucoma in each eye
* Requires IOP-lowering treatment in both eyes

Exclusion Criteria:

* Use of dorzolamide or carbonic anhydrase within 4 weeks
* Any other active ocular disease other than ocular hypertension or glaucoma (eg, uveitis, ocular infections or severe dry eye)
* Required chronic use of ocular medications other than study medication during the study (intermittent use of certain products eg, artificial tears are permitted)
* Use of oral, injectable or topical ophthalmic steroids within 21 days
* Any eye laser surgery within 3 months
* Any intraocular surgery (eg cataract surgery) within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Intraocular Pressure (IOP) | Baseline, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan